CLINICAL TRIAL: NCT01244828
Title: Long-term Study of Asenapine in Subjects With Residual Subtype, Receiving Multiple or/and High Dose Drugs, or Treatment Refractory Schizophrenia (Protocol P06238)
Brief Title: Long-term Study of Asenapine in Participants With Residual Subtype, Receiving Multiple or/and High Dose Drugs, or Treatment Refractory Schizophrenia (P06238)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06238; 132325 (Registry Identifier: Japic-CTI); MK-8274-042 (Other: Merck protocol number)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asenapine (Experimental): Asenapine 5 mg twice daily (BID) for the first week of treatment, then either 5 mg or 10 mg BID.
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Asenapine — 5 mg or 10 mg fast-dissolving sublingual tablets BID for up to 52 weeks

SUMMARY:
This is a multi-site, open-label fixed-flexible dose long-term study of asenapine in participants with schizophrenia. Participants in this study consist of schizophrenia with residual subtype or receiving high dose/multiple antipsychotic drugs, treatment refractory, or elderly participants with schizophrenia. The treatment period is up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 20 years
* Participants who meet at least one of the following:

  * current diagnosis of schizophrenia of residual subtype
  * received treatment with 3 or more antipsychotic drugs
  * treatment-refractory participants with schizophrenia
  * 65 years old and over with positive schizophrenia symptoms with score of 3 (mild) or more in 1 or more items in the positive subscale of the Positive and Negative Syndrome Scale (PANSS) at the baseline
* Participants who have a Clinical Global Impressions-Severity (CGI-S) score of at least 4 (moderately ill) at the baseline

Exclusion Criteria:

* Uncontrolled, unstable clinically significant medical condition
* Clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at Screening
* Positive pregnancy test at Screening, or the intention to become pregnant during the course of the study
* Seizure disorder beyond childhood (12 years old or younger)
* History of neuroleptic malignant syndrome
* Allergy or sensitivity to drugs such as psychotropics and antipsychotics
* Known history of or currently treated for narrow angle glaucoma
* Parkinson's disease
* Diagnosis of schizoaffective disorder; schizophreniform disorder
* Concurrent psychiatric disorder other than schizophrenia coded on Axis I; a primary diagnosis other than schizophrenia
* Diagnosis of borderline personality disorder
* Diagnosis of mental retardation or organic brain disorder
* Current (past 6 months) substance abuse or dependence according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria (excluding nicotine)
* Positive drug/alcohol tests at the Screening visit
* Imminent risk of self-harm or harm to others, in the Investigator's opinion
* Substance induced psychotic disorder or a behavioral disturbance thought to be due to substance abuse
* Currently under involuntary inpatient confinement
* Use of a non-approved drug in Japan within 12 weeks prior to informed consent
* Previously treated in an asenapine study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-04-05 (Actual); Primary Completion 2014-08-21 (Actual); Study Completion 2014-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine: All participants receive asenapine 5 mg twice daily (BID) for the first 7 days of treatment. After the initial 7-day period, the asenapine dose may be increased to 10 mg BID based on observed response to and toleration of the treatment. Asenapine dosing is flexible throughout the remainder of the study and may be adjusted, using the dose options of 5 and 10 mg BID, based on response and tolerability. The total duration of treatment is up to 52 weeks.
Period: Overall Study
Arm/Group | Asenapine
Started | 157 (Received study drug)
Completed | 79
Not Completed | 78
Not completed — Adverse Event | 37
Not completed — Withdrawal by Subject | 31
Not completed — Lack of Efficacy | 7
Not completed — Lost to Follow-up | 2
Not completed — Other reason (not specified) | 1

BASELINE CHARACTERISTICS:
Groups:
- Asenapine: All participants receive asenapine 5 mg BID for the first 7 days of treatment. After the initial 7-day period, the asenapine dose may be increased to 10 mg BID based on observed response to and toleration of the treatment. Asenapine dosing is flexible throughout the remainder of the study and may be adjusted, using the dose options of 5 and 10 mg BID, based on response and tolerability. The total duration of treatment is up to 52 weeks.
Arm/Group | Asenapine
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.37 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 81
Weight [Mean (Standard Deviation); unit: kg] | 59.45 (13.76)
Body Mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.04 (4.37)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] | 5.28 (0.47)
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] — For this measure, N=156
  mmol/L | 5.14 (0.74)
Insulin [Mean (Standard Deviation); unit: µIU/mL] | 6.35 (4.73)
Prolactin [Mean (Standard Deviation); unit: µg/L] | 43.92 (41.66)
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranged from 30 to 210 with a higher score indicating greater severity of symptoms.
  score on a scale | 89.99 (18.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight at Week 52
Description: For each participant, change from baseline in weight was calculated as the Week 52 value minus the baseline value.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Asenapine
Number analyzed (Participants) | 79
kg | 0.25 (5.23)

2. Primary Outcome: Change From Baseline in BMI at Week 52
Description: For each participant, change from baseline in BMI was calculated as the Week 52 value minus the baseline value.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Asenapine
Number analyzed (Participants) | 79
kg/m^2 | 0.07 (1.93)

3. Primary Outcome: Number of Participants With Extrapyramidal Symptoms
Description: This measure reports the overall number of participants with any of a group of adverse events that were defined to represent extrapyramidal symptoms. The number of participants with each of the individual adverse events within this definition is also presented, for terms that occurred in at least one participant. For this measure, all adverse event terms within the Medical Dictionary for Regulatory Activities (MedDRA) Standardized MedDRA Query (SMQ) for "extrapyramidal syndrome" were treated as extrapyramidal symptoms.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Asenapine
Number analyzed (Participants) | 157
participants
  Any extrapyramidal symptom | 24
  Restlessness | 3
  Akathisia | 3
  Dystonia | 2
  Extrapyramidal disorder | 10
  Parkinsonism | 1
  Tremor | 5
  Oculogyric crisis | 2
  Gait disturbance | 1

4. Primary Outcome: Change From Baseline in HbA1c at Week 52
Description: Blood samples for determination of HbA1c were obtained at baseline and during the study. For each participant, change from baseline in HbA1c at Week 52 was calculated as the Week 52 value minus the baseline value.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Asenapine
Number analyzed (Participants) | 79
percent | 0.00 (0.26)

5. Primary Outcome: Change From Baseline in Fasting Glucose at Week 52
Description: Blood samples for determination of fasting glucose level were obtained at baseline and during the study. For each participant, change from baseline in fasting glucose at Week 52 was calculated as the Week 52 level minus the baseline level.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Asenapine
Number analyzed (Participants) | 75
mmol/L | 0.11 (0.63)

6. Primary Outcome: Change From Baseline in Insulin at Week 52
Description: Blood samples for determination of insulin level were obtained at baseline and during the study. For each participant, change from baseline in insulin at Week 52 was calculated as the Week 52 level minus the baseline level.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Asenapine
Number analyzed (Participants) | 79
µIU/mL | 2.31 (11.93)

7. Primary Outcome: Change From Baseline in Prolactin at Week 52
Description: Blood samples for determination of prolactin level were obtained at baseline and during the study. For each participant, change from baseline in prolactin at Week 52 was calculated as the Week 52 level minus the baseline level.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 value of the measure.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Asenapine
Number analyzed (Participants) | 79
µg/L | 0.66 (24.20)

8. Primary Outcome: Change From Baseline in PANSS Total Score at Week 52
Description: The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was calculated as the sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Week 52 (calculated for a participant as Week 52 value minus baseline value); improvement in symptoms is represented by negative values.
Time Frame: Baseline and Week 52
Population: Participants who received at least one dose of study drug and had both a baseline and a Week 52 PANSS measurement.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 79
score on a scale | -11.08 (1.36)

9. Primary Outcome: Change From Baseline in PANSS Total Score at Final Assessment
Description: The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was calculated as the sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at the final assessment for a participant (calculated for a participant as final assessment value minus baseline value); improvement in symptoms is represented by negative values.
Time Frame: Baseline up to Week 52
Population: Participants who received at least one dose of study drug and had a baseline and at least one post-baseline PANSS measurement.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 153
score on a scale | -5.48 (1.08)

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 56 weeks)
Description: Analysis population is participants who received at least one dose of study drug.
Arm/Group | Asenapine
Serious Adverse Events (participants affected / at risk) | 14/157
Other Adverse Events (participants affected / at risk) | 111/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=157)
Pneumonia (Infections and infestations) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 4 (4)
Postresuscitation encephalopathy (Nervous system disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=157)
Constipation (Gastrointestinal disorders) | 10 (11)
Hypoaesthesia oral (Gastrointestinal disorders) | 17 (17)
Salivary hypersecretion (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 9 (9)
Pyrexia (General disorders) | 14 (17)
Nasopharyngitis (Infections and infestations) | 33 (63)
Contusion (Injury, poisoning and procedural complications) | 10 (12)
Fall (Injury, poisoning and procedural complications) | 10 (10)
Alanine aminotransferase increased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 11 (11)
Blood creatine phosphokinase increased (Investigations) | 10 (10)
Blood prolactin increased (Investigations) | 8 (8)
Weight decreased (Investigations) | 12 (12)
Weight increased (Investigations) | 20 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Extrapyramidal disorder (Nervous system disorders) | 10 (10)
Headache (Nervous system disorders) | 8 (9)
Somnolence (Nervous system disorders) | 20 (21)
Insomnia (Psychiatric disorders) | 8 (9)
Schizophrenia (Psychiatric disorders) | 17 (17)
Eczema (Skin and subcutaneous tissue disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Initial public presentation of the Investigator's results will occur only together with the other sites unless permission is obtained from Sponsor. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. In case of disagreement concerning appropriateness of materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues, prior to submission for publication/presentation.